CLINICAL TRIAL: NCT01595308
Title: A Pilot Study to Evaluate the Effect of Pomegranate Juice on Semen Parameters in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: POM Wonderful LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-002
Record Dates: First submitted 2012-04-04; First posted 2012-05-10 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Male Infertility
Keywords: Male infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomegranate juice (Experimental): Pomegranate juice
  Interventions: Dietary Supplement: Pomegranate juice

INTERVENTIONS:
Dietary Supplement: Pomegranate juice — Pomegranate juice

SUMMARY:
How daily consumption of pomegranate juice affects the concentration, morphology or motility of sperm in healthy men.

DETAILED DESCRIPTION:
To determine, in this pilot study, whether daily consumption of pomegranate juice (POM) affects the concentration, morphology or motility of sperm in healthy men. The purpose of the present pilot study is to examine the hypothesis that POM may improve semen parameters in men.

ELIGIBILITY:
Inclusion Criteria:

* 12 healthy men aged 18-40
* normal sperm counts

Exclusion Criteria:

* History of undescended testes or surgery to the scrotal contents,
* History of marijuana or alcohol abuse, hot tub usage at least 3 months prior to entry into the study
* No alpha adrenergic medications within two weeks of entry into the study,
* No anabolic steroid use,
* No anticholinergic or antimuscarinic drugs, use of colchicine, cimetidine, sulfasalazine, antipsychotics, antidepressants, immunosuppressive drugs prior use of any chemotherapeutic drugs, or UTI on screening visit.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
change in sperm counts | Baseline and 6 months
  The primary outcome will be change in sperm counts relative to baseline with and without POM.

SECONDARY OUTCOMES:
Change in Sperm count | 6 months
  The secondary outcome will be change in sperm counts relative to baseline with and without POM.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Rajfer, MD, Principal Investigator — Institute of Urologic Oncology at UCLA
Locations (1):
- Clinical Trials Program at University of California, Los Angeles, California, United States